CLINICAL TRIAL: NCT01776320
Title: A Phase 4, Open-Label, Non-Randomized, Clinical Trial to Evaluate the Efficacy, Safety and Satisfaction of VITAROS (Transdermal Topical Alprostadil) in Men With Erectile Dysfunction.
Brief Title: Efficacy, Safety and Satisfaction of VITAROS (Transdermal Topical Alprostadil) in Men With Erectile Dysfunction
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No medication
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Gerald Brock, Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103243
Record Dates: First submitted 2012-12-07; First posted 2013-01-28 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Topical Alprostadil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Alprostadil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VITAROS (Experimental): VITAROS (Alprostadil) 330 ug PRN (as needed) transdermal topical 4-8 weeks
  Interventions: Drug: Alprostadil

INTERVENTIONS:
Drug: Alprostadil — One unit of Vitaros(330ug of Alprostadil)once a week or once every two weeks for four or eight weeks.
  Other Names: VITAROS

SUMMARY:
A Phase 4 clinical trial that is open, with no blinding of subjects or randomization of treatment. Patients with erectile problems will be given the approved drug Vitaros to treat their condition. They will be given forms and questionnaires to complete. The information collected will be used to assess the effectiveness, safety and the satisfaction levels with this drug.

DETAILED DESCRIPTION:
Transdermal topical alprostadil has been approved for use in Canada as a treatment for erectile dysfunction. However, as this form of treatment is new, and Canada is the first country in the world to approve its use. There are very few published articles in literature to evaluate its clinical acceptance. By performing a Phase 4, Open-Label, Non-Randomized, Clinical Trial to Evaluate the Efficacy, Safety and Satisfaction of VITAROS (transdermal topical alprostadil) in Men with Erectile Dysfunction, this study can improve understanding of this method of treatment as compared to conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18y rs old and above
* Has mild-to-moderate erectile dysfunction
* Currently or previous treated for erectile dysfunction using PDE5 inhibitors, vacuum erection devices (VED), intra-cavernosal injections (ICI) and medical urethral system for erection (MUSE).
* Sexually active
* Has a regular sexual partner

Exclusion Criteria:

* Known allergy to alprostadil
* Unable to provide own informed consent
* Unable to understand and complete a questionnaire in English
* Unable to return for a post-treatment clinic evaluation
* Regular sexual partner is unable to understand and complete a questionnaire in English
* Sexual partner is a pregnant or lactating female

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of Topical alprostadil in the treatment of erectile dysfunction as measured by IIEF scores. | 4 - 8weeks

SECONDARY OUTCOMES:
Evaluate patient satisfaction of transdermal topical alprostadil when compared to patient's most current mode of therapy for erectile dysfunction. | 4 - 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Brock, MD, Principal Investigator — St.Joseph's Health Care
Locations (1):
- St. Joseph's Health Care London, London, Ontario, Canada

REFERENCES:
- [Background] Costa P, Potempa AJ. Intraurethral alprostadil for erectile dysfunction: a review of the literature. Drugs. 2012 Dec 3;72(17):2243-54. doi: 10.2165/11641380-000000000-00000. PMID 23170913